CLINICAL TRIAL: NCT04868240
Title: Effects of Concurrent Training on Metabolic Profile, Lung Function, Quality of Life and Stress in Sedentary Adults: A Randomized Controlled Trial
Brief Title: Concurrent Training and Metabolic Profile, Lung Function, Quality of Life and Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Fernanda Maria Antunes da Silva, MSc Fernanda Silva, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FCDEF UC (CIDAF); 2020.08759.BD (Other Grant/Funding Number: Fundação para a Ciência e a Tecnologia)
Record Dates: First submitted 2021-04-24; First posted 2021-04-30 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Sedentary Lifestyle; Metabolic Disorders; Concurrent Exercise; Lung Function Decreased; Stress; Quality of Life; Office Worker
MeSH Terms: conditions — Sedentary Behavior; Metabolic Diseases; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Single-blinded two-arm RCT with parallel-groups (1:1 allocation ratio).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concurrent Training Group (Experimental): The experimental group will perform 16-weeks of the concurrent training exercise.
  Interventions: Behavioral: Concurrent training program
- Control Group (No Intervention): Maintain their usual habits/activities, including not participate in any type of physical exercise.

INTERVENTIONS:
Behavioral: Concurrent training program — The experimental group will perform 16-weeks of exercise. The exercise sessions will occur three times/week.
  The participants should conduct their daily activities as usual outside of the study and maintain the same diet.
  Arms: Concurrent Training Group

SUMMARY:
Physical inactivity and sedentary time are highly prevalent worldwide and are associated with many adverse health outcomes. Workers adults spend two-thirds of their workday sitting, so they are particularly at risk. Exercise is considered a preventive and treatment tool for diseases, however, the effects of Concurrent Training (that is, aerobic plus resistance training) are not well established in healthy adults.

This research project aims to analyze the effects of a concurrent training program on metabolic profile, lung function, stress and quality of life, as well as body composition and physical fitness in sedentary adults.

This is a single-blinded two-arm RCT with parallel groups. After completion of baseline assessments, eligible participants will be randomized in a 1:1 ratio to participate in concurrent training group or control group. Repeat assessments will be taken immediately post 8 weeks and post 16 weeks of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with ages between 40 to 64 years old
* Physically inactive adults
* Full-time workers in a sedentary job
* BMI between 18 and 35 kg/m2
* Maintain the current diet and undergo all testing procedures

Exclusion Criteria:

* Chronic disease (e.g., diabetes, cardiovascular disease, pulmonary disease)
* Cognitive impairments and/or psychiatric conditions that could interfere with the study outcomes
* Take any medication that could interfere with the study outcomes
* Limitations that prevent them from practicing exercise
* History of heart failure/myocardial infarction
* Uncontrolled or abnormal blood pressure
* Smokers

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Lipid Profile at Week 16 | Baseline (Week 0) to follow-up (Week 16)
  The levels of total cholesterol, LDL-C, HDL-C, triglycerides, HbA1c, and glucose will be analyzed. These outcome measures have the same units of measure (mg/dL).
Change from Baseline in the Inflammatory Profile at Week 16 | Baseline (Week 0) to follow-up (Week 16)
  The cytokines IL-1β, IL-1ra, IL-10, IL-6, TNF-α, TGF-β, adiponectin and leptin will be analyzed. These outcome measures have the same units of measure (pg/ml).
Change from Baseline in the Fasting Insulin at Week 16 | Baseline (Week 0) to follow-up (Week 16)
  Insuline will be expressed in mU/L.
Change from Baseline in the Blood Pressure at Week 16 | Baseline (Week 0) to follow-up (Week 16)
  The systolic blood pressure (mmHg) and diastolic blood pressure (mmHg) will be measure through an automated oscillometric cuff.
Change from Baseline in Salivary Stress Hormones at Week 16 | Baseline (Week 0) to follow-up (Week 16)
  Salivary levels of cortisol, α-amylase, immunoglobulin A, and Lysozyme will be analyzed.
Change from Baseline in the Spirometric Values at Week 16 | Baseline (Week 0) to follow-up (Week 16)
  Spirometry will be performed to obtain the Forced Vital Capacity, Peak Expiratory Flow, and Forced Expiratory Volume in 1s.
  These outcome measures have the same units of measure, i.e., %predicted.
Change from Baseline in the "Satisfaction with Life" at Week 16 | Baseline (Week 0) to follow-up (Week 16)
  The "Satisfaction with Life Scale" questionnaire consists of 5-item formulated in the positive sense, that are answered using a 7-point Likert scale, where 1=strongly disagree and 7= strongly agree. Final scores range between 5 (low satisfaction) to 35 (high satisfaction).
Change from Baseline in the "Perceived Stress" at Week 16 | Baseline (Week 0) to follow-up (Week 16)
  The Perceived Stress Scale measures the perception of stress. Seven out of the 14-items are considered negative and seven as positive rated on a 5-point Likert scale. Final scores range between 0 to 56 points, with a higher score representing higher stress.
Change from Baseline in the "36-Item Short Form Survey (SF-36)" at Week 16 | Baseline (Week 0) to follow-up (Week 16)
  The 36-Item Short Form Survey is a generic instrument to evaluate health-related quality of life. SF-36 comprises 36 questions that cover 8 domains of health. Response choices for the items were on 2-, 3-, 5- or 6-point scales. Two-component scores are derived from 8 subdomains: a physical component (PC) and a mental component (MC). Higher scores on all subscales represent better health and functioning (>50).
Change from Baseline in the "World Health Organization Quality of Life Instruments - Bref" at Week 16 | Baseline (Week 0) to follow-up (Week 16)
  The World Health Organization Quality of Life Instruments - Bref, assesses the subjective quality of life and consists of 26 questions with responses on a 5-point Likert scale. Each domain is made up of questions where the scores vary between 1 and 5. The mean score in each domain represents the perception of the subject of their satisfaction with each aspect of quality of life. The higher the score, the better is their perception. There are no cut-points above or below which quality of life could be classified as "poor" or "good".

SECONDARY OUTCOMES:
Change from Baseline in the Body Composition at Week 16 | Baseline (Week 0) to follow-up (Week 16)
  Body weight (kg) and stature (cm) will be assessed to report BMI in kg/m^2. Values of skeletal muscle mass (kg) and fat mass (kg) will be determined using the tetrapolar bioimpedance (Inbody 270, USA).
Change from Baseline in the Cardiorespiratory Fitness at Week 16 | Baseline (Week 0) to follow-up (Week 16)
  Cardiorespiratory fitness will be assessed by the "Chester Step Test". The maximum test duration is 10 minutes (Level 5). VO2Max will be calculated by the CST software and expressed in mlso2/kg/min.
Change from Baseline in the Muscular Strength at Week 16 | Baseline (Week 0) to follow-up (Week 16)
  Handgrip strength will be measured by Jamar hand dynamometer. The test will be repeated twice with each hand. The score is the highest of the two readings (to the nearest kg).
Change from Baseline in the Flexibility at Week 16 | Baseline (Week 0) to follow-up (Week 16)
  Arms flexibility will be assessed by "Back Scratch test". Two attempts will be carried out on each side, and the result is the mean of the two measures.
  Legs flexibility will be assessed by "Modified Sit-and-reach test". Two measurements will be performed, and the result is the mean of the two measures.
Change from Baseline in the Levels of Physical Activity at Week 16 | Baseline (Week 0) to follow-up (Week 16)
  Sedentary time and physical activity levels (light, moderate and vigorous) will be assessed using a triaxial accelerometer (ActiGraph GT3X, US).
  These outcome measures have the same units of measure (min/day).

OTHER OUTCOMES:
Maximal Dynamic Strength (Estimated 1 RM) | Baseline (Week 0) to follow-up (Week 8)
  Experimental group participants will perform incremental loading tests to estimated 1 RM in free weights exercises.
Assessment of Dietary Intake | Baseline (Week 0) to follow-up (Week 16)
  Dietary habits will be assessed using a semi-quantitative Food Frequency Questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Fernanda Silva, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silva FM, Ferreira JP, Teixeira AM, Massart A, Duarte-Mendes P. Effects of combined aerobic-resistance training on health-related quality of life and stress in sedentary adults. Front Aging. 2025 Aug 18;6:1603635. doi: 10.3389/fragi.2025.1603635. eCollection 2025. PMID 40900743
- [Derived] Silva FM, Ferreira JP, Teixeira AM, Monteiro D, Duarte-Mendes P. The effect of smoking on lung function changes during a 16-week combined exercise program in middle-aged workers: a latent growth curve analysis. Eur J Appl Physiol. 2025 Nov;125(11):3223-3232. doi: 10.1007/s00421-025-05819-w. Epub 2025 May 31. PMID 40448859
- [Derived] Silva FM, Duarte-Mendes P, Ferreira JP, Carvalho E, Monteiro D, Massart A, Farinha C, Soares CM, Teixeira AM. Changes in Metabolic and Inflammatory Markers after a Combined Exercise Program in Workers: A Randomized Controlled Trial. Med Sci Sports Exerc. 2024 Nov 1;56(11):2156-2172. doi: 10.1249/MSS.0000000000003510. Epub 2024 Jun 27. PMID 38934517
- [Derived] Ferreira JP, Duarte-Mendes P, Teixeira AM, Silva FM. Effects of combined training on metabolic profile, lung function, stress and quality of life in sedentary adults: A study protocol for a randomized controlled trial. PLoS One. 2022 Feb 3;17(2):e0263455. doi: 10.1371/journal.pone.0263455. eCollection 2022. PMID 35113957